CLINICAL TRIAL: NCT00586482
Title: The Role of Nicotine Lozenges in Reducing Preoperative Exposure to Cigarette Smoke
Brief Title: Pilot Study: Preoperative Nicotine Lozenges
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, David Warner, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 06-002759
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Results first posted 2014-12-22 (Estimated); Last update posted 2014-12-22 (Estimated); Status verified 2014-12

CONDITIONS: Smoking
Keywords: cigarettes, surgery; Smokers scheduled for elective surgery
MeSH Terms: conditions — Smoking | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nicotine lozenge (Active Comparator): Nicotine lozenges, 2 or 4 mg, taken without restriction by mouth from 7 pm the evening before surgery until surgical admission the next day. Dosed according to time to first morning cigarette; if within 30 minutes of awakening, 4 mg lozenge used. If first cigarette smoked greater than 30 minutes of awakening, 2 mg lozenge used.
  Subjects also received an abstinence advisement: a brief (approximately 2 minute) behavioral intervention advising abstinence from smoking after 7 pm the night before surgery, the potential benefits of abstinence and to use a lozenge at usual smoking times.
  Interventions: Drug: Nicotine Lozenge; Behavioral: Abstinence Advisement
- Placebo lozenge (Placebo Comparator): Placebo lozenges, matching in appearance the 2 and 4 mg active nicotine lozenges, taken by mouth without restriction from 7 pm the night before surgery to the time of surgical admission the next day.
  Subjects also received an abstinence advisement: a brief (approximately 2 minute) behavioral intervention advising abstinence from smoking after 7 pm the night before surgery, the potential benefits of abstinence and to use a lozenge at usual smoking times.
  Interventions: Drug: Placebo Lozenge; Behavioral: Abstinence Advisement

INTERVENTIONS:
Drug: Nicotine Lozenge — Nicotine lozenges, 2 or 4 mg, taken without restriction by mouth from 7 pm the evening before surgery until surgical admission the next day and a 2 minute behavioral intervention. Dosed according to time to first morning cigarette; if within 30 minutes of awakening, 4 mg lozenge used. If first cigarette smoked greater than 30 minutes of awakening, 2 mg lozenge used.
  Other Names: Nicorette Lozenge
  Arms: Nicotine lozenge
Drug: Placebo Lozenge — Placebo lozenges, matching in appearance the 2 and 4 mg active nicotine lozenges, taken by mouth without restriction from 7 pm the night before surgery to the time of surgical admission the next day and a 2 minute behavioral intervention.
  Arms: Placebo lozenge
Behavioral: Abstinence Advisement — A brief (approximately 2 minute) behavioral intervention advising abstinence from smoking after 7 pm the night before surgery, the potential benefits of abstinence and to use a lozenge at usual smoking times.

SUMMARY:
The goal of this pilot study is to determine the feasibility and potential effect size of nicotine lozenges as an adjunct to maintain brief preoperative abstinence, defined as not smoking the day of surgery.

DETAILED DESCRIPTION:
Nicotine replacement therapy (NRT) helps patients maintain prolonged abstinence; whether it might also be efficacious in helping smokers maintain preoperative "fasting" from smoking is not known. A goal of this study is to determine how to best decrease smokers' exposure to cigarette smoke immediately before surgery. The specific aim of this study is to test the hypothesis that NRT in the form of nicotine lozenges will decrease the exposure to cigarette smoke prior to surgery. This is a randomized, double blinded, placebo controlled clinical trial examining the efficacy of the nicotine lozenge in increasing preoperative abstinence from cigarettes in patients scheduled for elective surgery. Current smokers scheduled for any of a wide variety of elective surgical procedures will be recruited in the Mayo Clinic Rochester Preoperative Evaluation Center. and will receive a brief practice-based intervention encouraging preoperative abstinence for at least 12 hours before admission to the surgical facility. They will be randomized to receive either active or placebo lozenge.

ELIGIBILITY:
Inclusion Criteria:

* Current cigarette smoker, defined as >100 cigarettes lifetime consumption and self report of smoking every day
* Scheduled for elective non-cardiac surgery

Exclusion Criteria:

* An inability to understand consent procedures
* History of an allergic reaction to nicotine replacement therapy
* History of sustained ventricular tachycardia
* Untreated hyperthyroidism or pheochromocytoma
* Currently utilizing pharmacologic agents specifically to treat nicotine dependence, including nicotine replacement therapy and bupropion (for a stop-smoking indication)
* Active (within the past 12 months) non-nicotine drug dependence
* Females who are pregnant or lactating
* Patients with phenylketonuria, because the lozenges contain aspartame, which is metabolized to phenylalanine.
* Lack of access to a telephone, as one follow-up will be performed using this means.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2006-08; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David O Warner, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Result] Warner DO, Kadimpati S. Nicotine lozenges to promote frief preopve abstinence from smoking: pilot study. Clin Health Promot 2(3):85-88, 2012.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from patients evaluated at the Mayo Clinic Pre-Operative Evaluation Center located in Rochester, Minnesota, in preparation for elective surgery.
Groups:
- Nicotine Lozenges: Nicotine lozenges, 2 or 4 mg, taken without restriction by mouth from 7 pm the evening before surgery until surgical admission the next day. Dosed according to time to first morning cigarette; if within 30 minutes of awakening, 4 mg lozenge used. If first cigarette smoked greater than 30 minutes of awakening, 2 mg lozenge used.
  Subjects also received an abstinence advisement: a brief (approximately 2 minute) behavioral intervention advising abstinence from smoking after 7 pm the night before surgery, the potential benefits of abstinence and to use a lozenge at usual smoking times.
Period: Overall Study
Arm/Group | Nicotine Lozenges | Placebo Lozenge
Started | 22 | 24
Completed | 22 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nicotine Lozenges | Placebo Lozenge | Total
Number analyzed (Participants) | 22 | 24 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.7 (14.0) | 49.8 (12.8) | 52.7 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 10 | 12 | 22
Region of Enrollment [Number; unit: participants]
  United States | 22 | 24 | 46
In-patient surgery [Number; unit: participants]
  In-Patient Elective Surgery | 12 | 13 | 25
  Out-Patient Elective Surgery | 10 | 11 | 21
Number of cigarettes per day [Mean (Standard Deviation); unit: Cigarettes per day] | 16.8 (6.7) | 17.9 (7.2) | 17.2 (7.0)
Fagerstrom Test for Nicotine Dependence [Mean (Standard Deviation); unit: Units on a scale] — This instrument consists of 6 questions related to cigarette smoking and nicotine dependency. Scores can range from 0 to 10. A score of 5 or less suggests low to moderate nicotine dependency. A score of 6 or higher indicates high nicotine dependency.
  Units on a scale | 6.7 (1.2) | 6.1 (1.4) | 6.4 (1.3)
Minnesota Nicotine Withdrawal Score [Mean (Standard Deviation); unit: units on a scale] — This item was measured using the Minnesota Nicotine Withdrawal Questionnaire, self-reported for the prior 24 hour period. This questionnaire consists of 15 items, each rated from 0 to 4, with a possible score of 0 to 60. A lower score indicates lesser withdrawal symptoms, and a higher score indicates greater withdrawal symptoms.
  units on a scale | 1.5 (0.9) | 1.5 (1.0) | 1.5 (1.0)
Pre-operative Abstinence Intention [Number; unit: participants]
  Intended to abstain prior to surgery | 18 | 19 | 37
  Did not intend to abstain prior to surgery | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Exhaled Carbon Monoxide Concentration
Time Frame: Morning of surgery, pre-operatively
Measure: Mean (Standard Deviation); unit: Parts per million
Arm/Group | Nicotine Lozenges | Placebo Lozenge
Number analyzed (Participants) | 22 | 24
Parts per million | 8.3 (7.5) | 12.7 (10.9)
Statistical Analysis 1: Comparison: Nicotine Lozenges vs Placebo Lozenge; A two-sided p value of less than or equal to 0.05 was considered statistically significant; Test type: Superiority or Other; p = 0.12, t-test, 2 sided

2. Secondary Outcome: Self-reported Abstinence
Description: Mean number who reported abstinence from smoking from the the time of baseline assessment until the morning of surgery.
Time Frame: Morning of surgery, pre-operatively
Measure: Number; unit: participants
Arm/Group | Nicotine Lozenges | Placebo Lozenge
Number analyzed (Participants) | 22 | 24
participants | 16 | 13
Statistical Analysis 1: Comparison: Nicotine Lozenges vs Placebo Lozenge; Test type: Superiority or Other; p = 0.23, Fisher Exact

3. Other Pre Specified Outcome: Self-reported Time to Last Cigarette
Time Frame: Morning of surgery, pre-operatively
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Nicotine Lozenges | Placebo Lozenge
Number analyzed (Participants) | 22 | 24
Hours | 21.8 (19.5) | 16.7 (11.3)
Statistical Analysis 1: Comparison: Nicotine Lozenges vs Placebo Lozenge; Test type: Superiority or Other; p = 0.29, t-test, 2 sided

4. Other Pre Specified Outcome: Minnesota Nicotine Withdrawal Score
Description: This item was measured using the Minnesota Nicotine Withdrawal Questionnaire, self-reported for the prior 24 hour period. This questionnaire consists of 15 items, each rated from 0 to 4, with a possible score of 0 to 60. A lower score indicates lesser withdrawal symptoms, and a higher score indicates greater withdrawal symptoms.
Time Frame: Morning of surgery, pre-operatively
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nicotine Lozenges | Placebo Lozenge
Number analyzed (Participants) | 22 | 24
units on a scale | 1.3 (1.0) | 1.4 (0.9)
Statistical Analysis 1: Comparison: Nicotine Lozenges vs Placebo Lozenge; Test type: Superiority or Other; p = 0.93, t-test, 2 sided

5. Other Pre Specified Outcome: Self-reported Abstinence From Smoking
Time Frame: Post-operative day 8
Measure: Number; unit: participants
Arm/Group | Nicotine Lozenges | Placebo Lozenge
Number analyzed (Participants) | 22 | 24
participants | 11 | 11
Statistical Analysis 1: Comparison: Nicotine Lozenges vs Placebo Lozenge; Test type: Superiority or Other; p = 1.0, Fisher Exact

ADVERSE EVENTS:
Arm/Group | Nicotine Lozenge | Placebo Lozenge
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/24
Other Adverse Events (participants affected / at risk) | 0/22 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No